CLINICAL TRIAL: NCT01271361
Title: Randomized Study to Assess the Effect of ThRombus Aspiration on Flow Area in STEMI Patients: an Optical Frequency Domain Imaging (OFDI) Study
Brief Title: Randomized Study to Assess the Effect of ThRombus Aspiration on Flow Area in STEMI Patients
Acronym: TROFI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T114E4
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; STEMI
Keywords: thrombus aspiration; Drug-Eluting Stent; optical frequency domain imaging (OFDI)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- primary PCI with thrombectomy (Experimental): thrombectomy before implantation of drug eluting stent
  Interventions: Procedure: primary PCI with thrombectomy
- primary PCI without thrombectomy (Active Comparator): implantation of a drug eluting stent without thrombectomy
  Interventions: Procedure: primary PCI without thrombectomy

INTERVENTIONS:
Procedure: primary PCI with thrombectomy — thrombectomy is performed before implantation of a drug eluting stent
  Other Names: Eliminate thrombectomy device; Nobori Biolimus A9 drug-eluting stent
  Arms: primary PCI with thrombectomy
Procedure: primary PCI without thrombectomy — no thrombectomy is performed before the implantation of a drug eluting stent
  Other Names: Nobori Biolimus A9 drug-eluting stent
  Arms: primary PCI without thrombectomy

SUMMARY:
The purpose of the study it to evaluate whether primary percutaneous coronary intervention (primary PCI) with a new thrombectomy device as compared to primary PCI without thrombectomy increases minimal flow area after stenting for treatment of patients presenting with ST-segment elevation myocardial infarction (STEMI) as assessed by OFDI.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention has been well established as the treatment of choice for the majority of patients presenting with acute ST elevation myocardial infarction (STEMI). However primary PCI alone is unable to remove intracoronary thrombus and this often results in distal embolisation, no reflow which in turn leads to impaired myocardial perfusion. This can result in left ventricular dysfunction and subsequently increased mortality.

The use of thrombectomy devices during percutaneous coronary intervention in the setting of acute ST elevation myocardial infarction has been recently shown to improve epicardial, myocardial perfusion, angiographical TIMI flow, blush score, or result in less embolisation. Moreover thrombus aspiration or rheolysis has been shown to decrease cardiac death and repeat myocardial infarction.

It is estimated that late stent malapposition is more common after stenting in the course of primary PCI as compared with elective PCI, and may predispose to stent thrombosis. Late malapposition may be related to underdeployment of stents at the time of primary PCI, and this may be due in part to thrombus behind the stent, which subsequently resolves and leads to stent malapposition. Removal of thrombus before stenting potentially could lead to better stent expansion and less late malapposition.

On the other hand, the impact of thrombus on acute and chronic luminal dimension is still unclear in a setting of primary PCI. After stenting, such thrombus either I) protrude into the lumen through the mesh of metallic stent struts or II) is crushed between the vessel wall and stent. Theoretically, the protruded thrombus can hinder the intra-luminal flow immediately after stenting, while the resorption of crushed thrombus against vessel wall might result at long term in stent malaposition.

Due to the limited ability of the conventional angiography and the intravascular ultrasound (IVUS) to detect thrombus, these aspects have not been investigated.

Optical coherence tomography has recently been shown to be feasible and to provide valuable information in the setting of acute myocardial infarction. This imaging modality has been shown to be even more sensitive to detect intraluminal mass (i.e. thrombus) and offers unique possibilities of analysis of coronary intervention in acute myocardial infarction.

TERUMO OFDI is a novel optical imaging device that uses a scanning laser as light source which centre wavelength is around 1.3 μm with sweeping range over 100 nm. The echo-time delay and the amplitude of light reflected from the tissue microstructure at different depths are determined by processing the interference between the tissue sample and a fixed reference mirror.

Compared to the conventional OCT imaging devices, OFDI has a higher temporal frame rate (160 frames/sec), with a faster pullback speed of maximally up to 40 mm/s. The safety and performance of the device has been investigated in the First-in-man study enrolling 19 patients where both IVUS and OFDI were performed. In the study, OFDI was associated with no device-related adverse events, and with a good correlation with IVUS measurement.

We hypothesize that TERUMO Eliminate® thrombectomy device will reduce the thrombus burden in STEMI patients and this will result in less intraluminal material and larger flow area, measured with OFDI. This will be clinically translated in a better restoration of blood flow and reduce further damage of the myocardium.

In addition, a reduction of thrombus burden would eventually result in less stent malaposition at 6 months. Given the benefits of reducing thrombus burden in STEMI as described above, the study may have important implications on the prove of the effectiveness of the thrombectomy device and the use of this imaging modality to assess its efficacy. To best assess benefits of thrombus removal, a randomized controlled study was considered the most appropriate method.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patients with a ST-elevation Myocardial Infarction documented in an ambulance or in a Cathlab with ≥2 mm ST segment elevation in at least two contiguous leads, presenting in the Cathlab <12 hours after the onset of symptoms lasting ≥20 min and having an angiographical visible stenosis (>30%) or TIMI≤ II in de-novo, native, previously unstented vessel.
* The single vessel coronary artery disease.
* Signed Informed Consent.
* The patient understands and accepts clinical follow-up and OFDI controls.
* Patients residence is in the area covered by hospital. Angiographic
* Vessel size should match available Nobori stent sizes (<4.0 mm, and >2.0 mm by visual assessment).

Additional Inclusion criteria (applicable only for France)

* Patients residence is in the area covered by hospital.
* Patient is affiliated to social security or equivalent system.

Exclusion Criteria:

* Pregnancy and women of child bearing potential (less than 50 years of age).
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, Biolimus A9, contrast material.
* Diameter Stenosis <30% in the target lesion.
* The multi-vessel coronary artery disease (DS>50%).
* Unprotected left main disease with a diameter stenosis of >30% by visual assessment.
* Distal vessel occlusion.
* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in sub-optimal imaging or excessive risk of complication from placement of an OFDI catheter.
* Fibrinolysis prior to PCI.
* Known thrombocytopaenia (PLT< 100,000/mm3).
* Contraindication to PCI, stenting, ASA, clopidogrel.
* Active bleeding or coagulopathy or patients at chronic anticoagulation therapy.
* Cardiogenic Shock.
* Significant comorbidities precluding clinical follow-up (as judged by investigators).
* Major planned surgery that requires discontinuation of dual antiplatelet therapy.
* Proximal RCA stenosis (>30%) if the infarct-related artery is mid-RCA or distal-RCA.
* People under judicial protection.
* A patient who has congenital heart disease, severe cardiac valve disorder and/or myocardial disease (excluding status post MI).
* Patient participating in other clinical research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
minimal flow area assessed by OFDI | at baseline procedure (post-stenting)
  Flow area is defined as: (Stent area + incomplete stent apposition area) - (intraluminal defect area attached to the wall + intraluminal defect area free from the wall)

SECONDARY OUTCOMES:
normalised minimal flow area | at baseline procedure (post stenting)
  defined as the ratio of minimal flow divided by stent area at the site of the minimal flow area
mean flow area/volume | at baseline procedure (post stenting) and at 6 months
intraluminal defect area/volume | at baseline procedure (post stenting) and at 6 months
mean stent area/volume | at baseline procedure (post stenting) and at 6 months
percent of malapposed struts | at baseline procedure (post stenting) and at 6 months
incomplete stent apposition (ISA) area/volume | at baseline procedure (post stenting) and at 6 months
percent of struts with coverage | at 6 months
healing index | at 6 months
tissues prolapse area/volume | at 6 months
procedure success | at baseline procedure
  attainment of <30% residual stenosis of the target lesion and no in-hospital target vessel failure
target vessel failure | at discharge, 1 month, 6 months and 12 months
  defined as cardiac death, reinfarction in the territory of infarction related vessel (Q wave and non-Q wave), or clinically driven target vessel revascularization - and its individual components
all-cause mortality | at discharge, 1 month, 6 months and 12 months
cardiac death, non-cardiovascular death, vascular death | at discharge, 1 month, 6 months and 12 months
any myocardial (re)infarction | at discharge, 1 month, 6 months and 12 months
target vessel revascularization | at discharge, 1 month, 6 months and 12 months
stent thrombosis according to ARC definition | at discharge, 1 month, 6 months and 12 months
other serious adverse events (SAEs) | at discharge, 1 month, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, Principal Investigator — Erasmus Medical Center, Rotterdam, Netherlands
Locations (5):
- Aarhus University Hospital Skejby, Aarhus, Denmark
- Clinique Pasteur, Toulouse, France
- Universität Leipzig - Herzzentrum, Leipzig, Germany
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - Maastad Hospital, Rotterdam

REFERENCES:
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Zijlstra F, Hoorntje JC, de Boer MJ, Reiffers S, Miedema K, Ottervanger JP, van 't Hof AW, Suryapranata H. Long-term benefit of primary angioplasty as compared with thrombolytic therapy for acute myocardial infarction. N Engl J Med. 1999 Nov 4;341(19):1413-9. doi: 10.1056/NEJM199911043411901. PMID 10547403
- [Background] Grines CL, Cox DA, Stone GW, Garcia E, Mattos LA, Giambartolomei A, Brodie BR, Madonna O, Eijgelshoven M, Lansky AJ, O'Neill WW, Morice MC. Coronary angioplasty with or without stent implantation for acute myocardial infarction. Stent Primary Angioplasty in Myocardial Infarction Study Group. N Engl J Med. 1999 Dec 23;341(26):1949-56. doi: 10.1056/NEJM199912233412601. PMID 10607811
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Sianos G, Papafaklis MI, Vaina S, Daemen J, van Mieghem CA, Van Domburg RT, Michalis LK, de Jaegere P, Serruys PW. Rheolytic thrombectomy in patients with ST-elevation myocardial infarction and large thrombus burden: the Thoraxcenter experience. J Invasive Cardiol. 2006 Jul;18 Suppl C:3C-7C. PMID 16883024
- [Background] Haeck JD, Koch KT, Bilodeau L, Van der Schaaf RJ, Henriques JP, Vis MM, Baan J Jr, Van der Wal AC, Piek JJ, Tijssen JG, Krucoff MW, De Winter RJ. Randomized comparison of primary percutaneous coronary intervention with combined proximal embolic protection and thrombus aspiration versus primary percutaneous coronary intervention alone in ST-segment elevation myocardial infarction: the PREPARE (PRoximal Embolic Protection in Acute myocardial infarction and Resolution of ST-Elevation) study. JACC Cardiovasc Interv. 2009 Oct;2(10):934-43. doi: 10.1016/j.jcin.2009.07.013. PMID 19850252
- [Background] Ikari Y, Sakurada M, Kozuma K, Kawano S, Katsuki T, Kimura K, Suzuki T, Yamashita T, Takizawa A, Misumi K, Hashimoto H, Isshiki T; VAMPIRE Investigators. Upfront thrombus aspiration in primary coronary intervention for patients with ST-segment elevation acute myocardial infarction: report of the VAMPIRE (VAcuuM asPIration thrombus REmoval) trial. JACC Cardiovasc Interv. 2008 Aug;1(4):424-31. doi: 10.1016/j.jcin.2008.06.004. PMID 19463340
- [Background] Vlaar PJ, Svilaas T, Vogelzang M, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan E, Suurmeijer AJ, Zijlstra F. A comparison of 2 thrombus aspiration devices with histopathological analysis of retrieved material in patients presenting with ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2008 Jun;1(3):258-64. doi: 10.1016/j.jcin.2008.03.014. PMID 19463309
- [Background] Sardella G, Mancone M, Bucciarelli-Ducci C, Agati L, Scardala R, Carbone I, Francone M, Di Roma A, Benedetti G, Conti G, Fedele F. Thrombus aspiration during primary percutaneous coronary intervention improves myocardial reperfusion and reduces infarct size: the EXPIRA (thrombectomy with export catheter in infarct-related artery during primary percutaneous coronary intervention) prospective, randomized trial. J Am Coll Cardiol. 2009 Jan 27;53(4):309-15. doi: 10.1016/j.jacc.2008.10.017. PMID 19161878
- [Background] Sardella G, Mancone M, Nguyen BL, De Luca L, Di Roma A, Colantonio R, Petrolini A, Conti G, Fedele F. The effect of thrombectomy on myocardial blush in primary angioplasty: the Randomized Evaluation of Thrombus Aspiration by two thrombectomy devices in acute Myocardial Infarction (RETAMI) trial. Catheter Cardiovasc Interv. 2008 Jan 1;71(1):84-91. doi: 10.1002/ccd.21312. PMID 17985382
- [Background] Silva-Orrego P, Colombo P, Bigi R, Gregori D, Delgado A, Salvade P, Oreglia J, Orrico P, de Biase A, Piccalo G, Bossi I, Klugmann S. Thrombus aspiration before primary angioplasty improves myocardial reperfusion in acute myocardial infarction: the DEAR-MI (Dethrombosis to Enhance Acute Reperfusion in Myocardial Infarction) study. J Am Coll Cardiol. 2006 Oct 17;48(8):1552-9. doi: 10.1016/j.jacc.2006.03.068. Epub 2006 Sep 26. PMID 17045887
- [Background] Svilaas T, van der Horst IC, Zijlstra F. Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS)--study design. Am Heart J. 2006 Mar;151(3):597.e1-597.e7. doi: 10.1016/j.ahj.2005.11.010. PMID 16504620
- [Background] Burzotta F, Trani C, Romagnoli E, Mazzari MA, Rebuzzi AG, De Vita M, Garramone B, Giannico F, Niccoli G, Biondi-Zoccai GG, Schiavoni G, Mongiardo R, Crea F. Manual thrombus-aspiration improves myocardial reperfusion: the randomized evaluation of the effect of mechanical reduction of distal embolization by thrombus-aspiration in primary and rescue angioplasty (REMEDIA) trial. J Am Coll Cardiol. 2005 Jul 19;46(2):371-6. doi: 10.1016/j.jacc.2005.04.057. PMID 16022970
- [Background] De Luca G, Dudek D, Sardella G, Marino P, Chevalier B, Zijlstra F. Adjunctive manual thrombectomy improves myocardial perfusion and mortality in patients undergoing primary percutaneous coronary intervention for ST-elevation myocardial infarction: a meta-analysis of randomized trials. Eur Heart J. 2008 Dec;29(24):3002-10. doi: 10.1093/eurheartj/ehn389. Epub 2008 Sep 5. PMID 18775918
- [Background] Chevalier B, Gilard M, Lang I, Commeau P, Roosen J, Hanssen M, Lefevre T, Carrie D, Bartorelli A, Montalescot G, Parikh K. Systematic primary aspiration in acute myocardial percutaneous intervention: a multicentre randomised controlled trial of the export aspiration catheter. EuroIntervention. 2008 Aug;4(2):222-8. doi: 10.4244/eijv4i2a40. PMID 19110787
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet. 2008 Jun 7;371(9628):1915-20. doi: 10.1016/S0140-6736(08)60833-8. PMID 18539223
- [Background] Kubo T, Imanishi T, Takarada S, Kuroi A, Ueno S, Yamano T, Tanimoto T, Matsuo Y, Masho T, Kitabata H, Tsuda K, Tomobuchi Y, Akasaka T. Assessment of culprit lesion morphology in acute myocardial infarction: ability of optical coherence tomography compared with intravascular ultrasound and coronary angioscopy. J Am Coll Cardiol. 2007 Sep 4;50(10):933-9. doi: 10.1016/j.jacc.2007.04.082. Epub 2007 Aug 20. PMID 17765119
- [Background] Gonzalo N, Barlis P, Serruys PW, Garcia-Garcia HM, Onuma Y, Ligthart J, Regar E. Incomplete stent apposition and delayed tissue coverage are more frequent in drug-eluting stents implanted during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction than in drug-eluting stents implanted for stable/unstable angina: insights from optical coherence tomography. JACC Cardiovasc Interv. 2009 May;2(5):445-52. doi: 10.1016/j.jcin.2009.01.012. PMID 19463469
- [Background] Hara H, Nakamura M, Komatsu H, Ikeda N, Shinji H, Makino K, Itaya H, Yamamoto M, Itou N, Tsunoda T, Sugi K. Comparison of the in vitro performance of 6 and 7 French aspiration catheters. EuroIntervention. 2007 Feb;2(4):487-92. PMID 19755289
- [Background] Grayson AD, Moore RK, Jackson M, Rathore S, Sastry S, Gray TP, Schofield I, Chauhan A, Ordoubadi FF, Prendergast B, Stables RH; North West Quality Improvement Programme in Cardiac Interventions. Multivariate prediction of major adverse cardiac events after 9914 percutaneous coronary interventions in the north west of England. Heart. 2006 May;92(5):658-63. doi: 10.1136/hrt.2005.066415. Epub 2005 Sep 13. PMID 16159983
- [Background] Guedes A, Keller PF, L'Allier PL, Lesperance J, Gregoire J, Tardif JC. Long-term safety of intravascular ultrasound in nontransplant, nonintervened, atherosclerotic coronary arteries. J Am Coll Cardiol. 2005 Feb 15;45(4):559-64. doi: 10.1016/j.jacc.2004.10.063. PMID 15708704
- [Background] Johansson P, Lunden M, Ekstrom L, Grip L, Wennerblom B. Intensive use of intravascular ultrasound during coronary angioplasty. A six-month campaign. Scand Cardiovasc J. 2001 Mar;35(2):75-9. doi: 10.1080/140174301750164655. PMID 11405500
- [Background] Vranckx P, Cutlip DE, Mehran R, Kint PP, Silber S, Windecker S, Serruys PW. Myocardial infarction adjudication in contemporary all-comer stent trials: balancing sensitivity and specificity. Addendum to the historical MI definitions used in stent studies. EuroIntervention. 2010 Feb;5(7):871-4. doi: 10.4244/eijv5i7a146. No abstract available. PMID 20142206
- [Derived] Muramatsu T, Garcia-Garcia HM, Onuma Y, Zhang YJ, Bourantas CV, Diletti R, Iqbal J, Radu MD, Ozaki Y, Serruys PW; TROFI investigators. Intimal flaps detected by optical frequency domain imaging in the proximal segments of native coronary arteries: an innocent bystander? Insights from the TROFI Trial. Circ J. 2013;77(9):2327-33. doi: 10.1253/circj.cj-13-0357. Epub 2013 Jun 15. PMID 23979567
- [Derived] Muramatsu T, Garcia-Garcia HM, Onuma Y, Zhang YJ, Bourantas CV, Diletti R, Iqbal J, Radu MD, Ozaki Y, Serruys PW; on behalf of the TROFI investigators. Intimal Flaps Detected by Optical Frequency Domain Imaging in the Proximal Segments of Native Coronary Arteries. Circ J. 2013 Jun 15. Online ahead of print. PMID 23778184
- [Derived] Muramatsu T, Garcia-Garcia HM, Lee IS, Bruining N, Onuma Y, Serruys PW. Quantitative optical frequency domain imaging assessment of in-stent structures in patients with ST-segment elevation myocardial infarction: impact of imaging sampling rate. Circ J. 2012;76(12):2822-31. doi: 10.1253/circj.cj-12-0536. Epub 2012 Aug 29. PMID 22971949